CLINICAL TRIAL: NCT03192670
Title: A Study of Low-level Light Therapy Using Photo-activated Modulation Ameliorates Cognitive Deficits by Enhancing Cerebral Blow Flow
Brief Title: A Study of Low-level Light Therapy Using Photo-activated Modulation Ameliorates Cognitive Deficits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yong-il Shin, MD (Other)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Sponsor-Investigator, Yong-il Shin, MD, Professor, Pusan National University
Organization: Pusan National University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNUYH-03-2017-003, SMC-2016-1
Record Dates: First submitted 2017-06-08; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Mild Cognitive Impairment; Cerebral Blood Flow; Low-level Light Therapy; Brain Activity
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sham control group (Sham Comparator): Sham control group received same procedure without LED-T. Device: Low-level light therapy device approved by the ethics committees of Pusan National hospital and conformity MSDS as safe treatment device for brain diseases Parameters: Neuroimaging assessment(fMRI, SPECT), Neuropsychological Behavioral Assessment(SNSB, K-MoCA, Corsiblock test, K-MBI, K-ADL, GDS, EQ-5D)
  Interventions: Device: Low-level light therapy device
- CA(Carotid artery)-stimulation group (Experimental): In CA group, total sessions of the LED-T was done for each groups and assessment of parameters was followed that.
  Each group subject underwent LED therapy (30 min) once a day for 20 days, commencing at Baseline screening test.
  Device: Low-level light therapy device approved by the ethics committees of Pusan National hospital and conformity MSDS as safe treatment device for brain diseases Parameters: Neuroimaging assessment(fMRI, SPECT), Neuropsychological Behavioral Assessment(SNSB, K-MoCA, Corsiblock test, K-MBI, K-ADL, GDS, EQ-5D)
  Interventions: Device: Low-level light therapy device
- VA(Vertebral artery)-stimulation group (Experimental): In VA group, total sessions of the LED-T was done for each groups and assessment of parameters was followed that.
  Each group subject underwent LED therapy (30 min) once a day for 20 days, commencing at Baseline screening test.
  Device: Low-level light therapy device approved by the ethics committees of Pusan National hospital and conformity MSDS as safe treatment device for brain diseases Parameters: Neuroimaging assessment(fMRI, SPECT), Neuropsychological Behavioral Assessment(SNSB, K-MoCA, Corsiblock test, K-MBI, K-ADL, GDS, EQ-5D)
  Interventions: Device: Low-level light therapy device
- CA+VA dual stimulation group (Experimental): In CA+VA group, total sessions of the LED-T was done for each groups and assessment of parameters was followed that.
  Each group subject underwent LED therapy (30 min) once a day for 20 days, commencing at Baseline screening test.
  Device: Low-level light therapy device approved by the ethics committees of Pusan National hospital and conformity MSDS as safe treatment device for brain diseases Parameters: Neuroimaging assessment(fMRI, SPECT), Neuropsychological Behavioral Assessment(SNSB, K-MoCA, Corsiblock test, K-MBI, K-ADL, GDS, EQ-5D)
  Interventions: Device: Low-level light therapy device

INTERVENTIONS:
Device: Low-level light therapy device — Peak wavelength:610nm, Power intensity: 1.7mW/cm2, Energy density: 2.0J/cm2, Skin-adhesive light-emitting probes: spot size, 1cm diameter

SUMMARY:
The primary objective of this study is to confirm and compare the effect of methods of Low-level light therapy (LED-T) in the mild cognitive impairment.

DETAILED DESCRIPTION:
Total 168 patients were recruited and randomized to receive either real or sham-LED-T. Real experimental groups were divided into three groups; CA group, VA group, CA+VA dual group. Each group received LED-T (30 min) once a day for 30 days. Each groups LED-T positioned at following locations;

* CA group on the superior border of the thyroid cartilage, and anterior to the sternocleidomastoid muscle based on Korea traditional therapy called Inyoung(ST9)
* VA group on the upper abdomen, spinous process of the 2nd cervical vertebra upper margin based on Korea traditional therapy called CunChu
* CA+VA dual group on the CA position (ST9), and VA position (BL10) The patients were initially evaluated at baseline, immediately, 4wks after intervention.

Study type : Interventional Study Phase : Not provided Study Design : Allocation : Randomized Intervention Model : Parallel Assignment Masking : Single Blind (Investigator) Primary Purpose : Treatment, intervention Condition : Mild cognitive impairment, Health subjects

Intervention :

* Low-level light therapy device (Peak wavelength:610nm, Power intensity: 1.7mW/cm2, Energy density: 2.0J/cm2, Skin-adhesive light-emitting probes: spot size, 1cm diameter),
* Parameters : Neuroimaging assessement: fMRI, SPECT, Neuropsychological behavioral assessment: SNSB; Seoul Neuropsychological screening battery, K-MoCA, Corsi-block test, K-MBI, K-ADL, GDS, EQ-5D, Neurophysiological assessment: MEP, Motor evoked potential, Gene test(BNDF, ApoE)

Study Arms

* Experimental : Sham control group and real stimulation group.
* In each group, total sessions of the Low-level light therapy (LED-T) was done for intervention was followed after that.
* Subjects received LED-T (30 min) once a day for 30 days.
* The sham control group was kept without LED-T

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ages older than 55 years old
2. Subjects who has K-MoCA assessment score less than 23
3. Subjects who understand the purpose of the study and acquired the consent of the subjects or caregiver

Exclusion Criteria:

1. Subjects who have K-MMSE less than 19
2. Subjects who have pre-existing and present-existing neurological diseases as CNS lesion
3. Subjects who have psychiatric disease such as depression, schizophrenia, bipolar disease, or dementia
4. Subjects who is estimated as not appropriate for the study by the investigators

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2017-06-20 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological Behavioral Assessment 1 | Baseline, Change from Baseline SNSB at immediately after intervention , Change from Baseline SNSB at 4 weeks after intervention
  SNSB

SECONDARY OUTCOMES:
Neuropsychological Behavioral Assessment 2 | Baseline, Change from Baseline Corsi-block test at immediately after intervention , Change from Baseline Corsi-block test at 4 weeks after intervention
  Corsi-block test
Neuropsychological Behavioral Assessment 3 | Baseline, Change from Baseline K-MoCA at immediately after intervention , Change from Baseline K-MoCA at 4 weeks after intervention
  K-MoCA
ADL assessment 1 | Baseline, Change from Baseline K-MBI at immediately after intervention , Change from Baseline K-MBI at 4 weeks after intervention
  K-MBI
ADL assessment 2 | Baseline, Change from Baseline K-ADL at immediately after intervention , Change from Baseline K-ADL at 4 weeks after intervention
  K-ADL
Depression assessment | Baseline, Change from Baseline GDS-SF at immediately after intervention , Change from Baseline GDS-SF at 4 weeks after intervention
  GDS-SF
Quality of Life assessment | Baseline, Change from Baseline EQ-5D at immediately after intervention , Change from Baseline EQ-5D at 4 weeks after intervention
  EQ-5D
Gene test 1 | Baseline, Change from Baseline BNDF at immediately after intervention , Change from Baseline BNDF at 4 weeks after intervention
  BNDF
Gene test 2 | Baseline, Change from Baseline ApoE at immediately after intervention , Change from Baseline ApoE at 4 weeks after intervention
  ApoE
Neuroimaging Assessment 1 | Baseline, Change from Baseline fMRI at immediately after intervention , Change from Baseline fMRI at 4 weeks after intervention
  fMRI
Neuroimaging Assessment 2 | Baseline, Change from Baseline SPECT at immediately after intervention , Change from Baseline SPECT at 4 weeks after intervention
  SPECT

CONTACTS AND LOCATIONS:
Overall Officials: Yong-il Shin, M.D, Ph.D, Study Chair — Pusan National University Yangsan Hospital
Locations (2):
- South Korea (2):
  - Pusan National University Yangsan Hospital Yangsan, Yangsan, Gyeongsangnam-do
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee HI, Lee SW, Kim NG, Park KJ, Choi BT, Shin YI, Shin HK. Low-level light emitting diode therapy promotes long-term functional recovery after experimental stroke in mice. J Biophotonics. 2017 Dec;10(12):1761-1771. doi: 10.1002/jbio.201700038. Epub 2017 May 2. PMID 28464523
- [Background] Lee HI, Lee SW, Kim SY, Kim NG, Park KJ, Choi BT, Shin YI, Shin HK. Pretreatment with light-emitting diode therapy reduces ischemic brain injury in mice through endothelial nitric oxide synthase-dependent mechanisms. Biochem Biophys Res Commun. 2017 May 13;486(4):945-950. doi: 10.1016/j.bbrc.2017.03.131. Epub 2017 Mar 24. PMID 28347821
- [Background] Lee HI, Lee SW, Kim NG, Park KJ, Choi BT, Shin YI, Shin HK. Low-level light emitting diode (LED) therapy suppresses inflammasome-mediated brain damage in experimental ischemic stroke. J Biophotonics. 2017 Nov;10(11):1502-1513. doi: 10.1002/jbio.201600244. Epub 2017 Feb 6. PMID 28164443
- [Background] Lee HI, Park JH, Park MY, Kim NG, Park KJ, Choi BT, Shin YI, Shin HK. Pre-conditioning with transcranial low-level light therapy reduces neuroinflammation and protects blood-brain barrier after focal cerebral ischemia in mice. Restor Neurol Neurosci. 2016;34(2):201-14. doi: 10.3233/RNN-150559. PMID 26889965
- [Background] Hong GY, Shin BC, Park SN, Gu YH, Kim NG, Park KJ, Kim SY, Shin YI. Randomized controlled trial of the efficacy and safety of self-adhesive low-level light therapy in women with primary dysmenorrhea. Int J Gynaecol Obstet. 2016 Apr;133(1):37-42. doi: 10.1016/j.ijgo.2015.08.004. Epub 2015 Dec 2. PMID 26797192